CLINICAL TRIAL: NCT04042402
Title: An Open-Label Roll-Over Study to Evaluate the Long-Term Safety and Efficacy of DCR-PHXC Solution for Injection (Subcutaneous Use) in Patients With Primary Hyperoxaluria
Brief Title: Long Term Extension Study in Patients With Primary Hyperoxaluria
Acronym: PHYOX3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCR-PHXC-301
Record Dates: First submitted 2019-07-10; First posted 2019-08-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1); Primary Hyperoxaluria Type 2 (PH2); Kidney Diseases; Urologic Diseases; Genetic Disease; Primary Hyperoxaluria Type 3 (PH3)
Keywords: Primary Hyperoxaluria; PH1; PH2; RNAi; GalNAc; LDHA; LDH; siRNA; PH3
MeSH Terms: conditions — Primary hyperoxaluria type 1; Primary hyperoxaluria type 2; Kidney Diseases; Urologic Diseases; Genetic Diseases, Inborn; Hyperoxaluria, Primary | interventions — nedosiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label (Experimental): Open label, monthly subcutaneous injection
  Interventions: Drug: DCR-PHXC

INTERVENTIONS:
Drug: DCR-PHXC — Multiple fixed doses of DCR-PHXC by subcutaneous (SC) injection
  Other Names: Nedosiran

SUMMARY:
The proposed study is designed to provide patients previously enrolled in Phase 1 and 2 studies of DCR-PHXC and their siblings (<18 years old) long-term access to DCR-PHXC, and to evaluate the long-term safety and efficacy of DCR-PHXC in patients with PH.

ELIGIBILITY:
Key Inclusion Criteria:

•Participant successfully completed a Dicerna Pharmaceuticals, Inc. study of DCR PHXC.

OR Participant is the sibling of a participant who successfully completed a Dicerna Pharmaceuticals, Inc. study of DCR PHXC. Siblings must be younger than 18 years of age and must have genetically confirmed PH.

* For participants rolling over from a multidose study of DCR-PHXC, enrollment should occur within a window of 25 to 75 days from the last dose of study intervention.
* Estimated GFR at screening ≥ 30 mL/min normalized to 1.73 m2 body surface area (BSA), calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) formula in participants aged ≥ 18 years, or the multivariate equation by Schwartz in participants aged 12 months to 17 years. In Japan, the cystatin C-based Uemura formula will be used for participants aged 12 months to <2 years, the creatinine-based Uemura formula by will be used for participants aged 2 to 17 years, and the equation by Matsuo will be used in participants aged ≥ 18 years.

Key Exclusion Criteria:

* Renal or hepatic transplantation (prior or planned within the study period)
* Plasma oxalate > 30 µmol/L
* Currently on dialysis
* Documented evidence of clinical manifestations of systemic oxalosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
The annual rate of decline in eGFR in participants with PH1 | Annual change from baseline
  To evaluate the effect of DCR PHXC on estimated glomerular filtration rate (eGFR) in participants with PH1

SECONDARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAE) and SAEs associated with abnormal 12 lead electrocardiogram (ECG) readings | TEAEs and SAEs are evaluated monthly for 6 years
  To evaluate the safety and tolerability of DCR PHXC when administered monthly to patients with primary hyperoxaluria (PH) via change from baseline and abnormal ECG findings.
  Standard 12-lead ECGs will be performed in the supine position after the subject has rested comfortably for 10 minutes. The parameters assessed will be rhythm, ventricular rate, PR interval, QRS duration, QT interval, and corrected QT interval (QTcF, Fridericia correction). The Investigator or designee is responsible for reviewing the ECG(s) to assess whether the results are within normal limits and to determine the clinical significance of the results.
  Standardized ECG acquisition equipment will be provided to all clinical trial sites at the start of the trial, to ensure parity across all sites.
The incidence and severity of treatment-emergent adverse events (TEAE) and SAEs associated with abnormal physical examination findings | TEAEs and SAEs are evaluated monthly for 6 years
  To evaluate the safety and tolerability of DCR PHXC when administered monthly to patients with primary hyperoxaluria (PH) via change from baseline and incidence of abnormal physical exam findings.
  A full physical examination will include a complete review of body systems: eyes, ears, nose, and throat, chest/respiratory, heart/cardiovascular, gastrointestinal/liver, musculoskeletal/extremities, dermatological/skin, thyroid/neck, lymph nodes, and neurological. A full physical exam is done at Screening, Day 180 and if a participant ends the study early.
  A brief physical examination will minimally include chest/respiratory, heart/cardiovascular, dermatological/skin, and gastrointestinal/liver. A brief physical examination will be performed at the Investigator's discretion at all other visits.
The incidence and severity of treatment-emergent adverse events (TEAE) and SAEs associated with abnormal vital signs | TEAEs and SAEs are evaluated monthly for 6 years
  To evaluate the safety and tolerability of DCR PHXC when administered monthly to patients with primary hyperoxaluria (PH) via the change from baseline and incidence of abnormal vital signs.
  Vital signs include blood pressure, pulse/heart rate, oral body temperature, and respiratory rate.
  Parameters will be measured in the supine position, using an automated instrument or manually, after the participant has rested comfortably for 10 minutes. In the pediatric population, an age-appropriate cuff size should be used for blood pressure measurements.
  Temperature will be obtained in degrees Celsius (°C), pulse rate will be counted for a full minute and recorded in beats per minute, and respirations will be counted for a full minute and recorded in breaths per minute.
The incidence and severity of treatment-emergent adverse events (TEAE) and SAEs related to abnormal clinical laboratory tests (hematology, chemistry, coagulation parameters, and urinalysis) | TEAEs and SAEs are evaluated monthly for 6 years
  To evaluate the safety and tolerability of DCR PHXC when administered monthly to patients with primary hyperoxaluria (PH) via the change from baseline and incidence of abnormal clinical laboratory tests.
To identify the proportion of participants with normalized or near-normalized 24 hour urinary oxalate (Uox) | 24 hour urine collections (if applicable) are performed monthly for 6 months (or quarterly for PH1 multidose rollovers), quarterly for 2 1/2 years (or monthly for PH2/PH3 multidose rollovers until Month 12), and every 6 months for 3 years after that.
  The proportion of participants with a 24 hour Uox level (< 0.46 mmol/24 hours or ≥ 0.46 - < 0.60 mmol/24 hours [adjusted per 1.73 m2 body surface area (BSA) in participants aged < 18 years]) at each assessment time point throughout the study in PH1, PH2, and PH3 participant subgroups
To identify the percentage of participants with spot urinary oxalate-to-creatinine ratio ≤ the ULN or ≤ 1.5 x ULN | Spot urine collections are performed monthly for 6 months (or quarterly for PH1 multidose rollovers), quarterly for 2 1/2 years (or monthly for PH2/PH3 multidose rollovers until Month 12), and every 6 months for 3 years after that.
  The percentage of participants with spot urinary oxalate-to-creatinine ratio ≤ the ULN or ≤ 1.5 x ULN at each assessment time point throughout the study in PH1, PH2, and PH3 participant subgroups
To assess the effect of DCR-PHXC on stone events in patients with PH | Evaluated yearly for 6 years
  Change from Baseline in the number of stone events over a 12-month period, annually in Year 1, Year 2, etc. in PH1, PH2, and PH3 participant subgroups
To assess the effect of DCR-PHXC on stone burden grade in patients with PH | Evaluated yearly for 6 years
  Change from Baseline in the stone burden grade at Year 1, Year 2, etc. in PH1, PH2, and PH3 participant subgroups
To assess the effect of DCR-PHXC in nephrocalcinosis grade in patients with PH | Evaluated yearly for 6 years
  Change from Baseline in nephrocalcinosis grade at Year 1, Year 2, etc. in PH1, PH2, and PH3 participant subgroups
To evaluate the incidence of chronic kidney disease (CKD) and end-stage renal disease (ESRD) in participants with PH | eGFR is evaluated monthly for 6 months (or quarterly for multidose rollovers), quarterly for 2 1/2 years, and every 6 months for 3 years after that.
  The number of participants with severe CKD (GFR = 15-29 mL/min) or ESRD (GFR <15 mL/min); adjusted per 1.73 m2 BSA in participants aged < 18 years in PH1, PH2, and PH3 participant subgroups
Change from Baseline in the Short Form (36) Health Survey (SF-36®) in PH1, PH2, and PH3 participant subgroups | Surveys are administered at screening, Day 180, yearly for 3.5 years, then at Month 72 (EOS).
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The SF 36 is a set of generic, coherent, and easily administered quality-of-life measures that taps 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The 36 items are identical to the MOS SF 36 described in Ware and Sherbourne (1992). Participants respond to each item on a categorical scale. Categorical answers are transformed to a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Change from Baseline in the EQ-5D-5L™ in adults in PH1, PH2, and PH3 participant subgroups | Surveys are administered at screening, Day 180, yearly for 3.5 years, then at Month 72 (EOS).
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The EQ-5D-5L consists of the EQ 5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the 5 dimensions can be combined into a 5-digit number that describes the participant's health state.
  The EQ VAS records the participant's self-rated health on a 20-cm vertical VAS, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine.' Participants are asked to place an "X" on the line that represents their health on that day.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL™) in children in PH1, PH2, and PH3 participant subgroups | Surveys are administered at screening, Day 180, yearly for 3.5 years, then at Month 72 (EOS).
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The 23-item PedsQL is comprised of 5 items in the Emotional, Social, and School Functioning dimensions (Psychosocial Health) and 8 items in the Physical Functioning (Physical Health) dimension. Items are reverse-scored on a 0 to 4 Likert scale and linearly transformed to a 0 to 100 scale, so that higher scores indicate better functioning and HRQOL. Scale Scores are the sum of the items in each dimension, divided by the number of items answered.
To assess the efficacy of DCR PHXC in reducing Uox burden in patients with PH: TWS AUC | Monthly for 4 months (D90 through D180)
  Time-weighted standardized area under the curve (TWS AUC) of 24-hour Uox from Day 90 to Day 180, based on percent change from Baseline in PH1, PH2, and PH3 participant subgroups. This endpoint will only be assessed in participants previously randomized to placebo in a previous study of DCR- PHXC and pediatric siblings.
To assess the long-term efficacy of DCR PHXC in reducing Uox burden in patients with PH | 24 hour urine collections (if applicable) are performed monthly for 6 months (or quarterly for PH1 multidose rollovers), quarterly for 2 1/2 years (or monthly for PH2/PH3 multidose rollovers until Month 12), and every 6 months for 3 years after that.
  Percent change from Baseline in 24-hour Uox at each assessment time point throughout the study in PH1, PH2, and PH3 participant subgroups. In those participants randomized to placebo in a previous study of DCR-PHXC and pediatric siblings, this endpoint will be assessed only after Month 6
To assess the long-term efficacy of DCR-PHXC in reducing Uox burden in patients with PH | Spot urine collections are performed monthly for 6 months (or quarterly for PH1 multidose rollovers), quarterly for 2 1/2 years (or monthly for PH2/PH3 multidose rollovers until Month 12), and every 6 months for 3 years after that.
  Percent and absolute change from Baseline in spot urinary oxalate-to-creatinine ratio at each assessment time point throughout the study in PH1, PH2, and PH3 participant subgroups. In pediatric siblings, this endpoint will be assessed only after Month 6

OTHER OUTCOMES:
To evaluate the effect of DCR PHXC on eGFR in participants with PH2 and PH3 | Annual change from baseline
  The annual rate of decline in eGFR in participants with PH2 and PH3
To characterize the PK of DCR PHXC in patients with PH by observing minimum concentration (Cmin). | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including minimum observed concentration (Cmin)
To characterize the PK of DCR PHXC in patients with PH by observing maximum concentration (Tmax). | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including time to maximum concentration (Tmax)
To characterize the PK of DCR PHXC in patients with PH by observing terminal elimination half-life (t1/2). | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including terminal elimination half-life (t1/2)
To characterize the PK of DCR PHXC in patients with PH by observing clearance. | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including clearance (CL)
To characterize the PK of DCR PHXC in patients with PH by observing volume of distribution of estimates. | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including volume of distribution (V) estimates
To characterize the PK of DCR PHXC in patients with PH by observing the area under the curve (AUC) | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including secondary parameters of area under the curve (AUC)
To characterize the PK of DCR PHXC in patients with PH by observing maximum observed concentration (Cmax). | Participants rolling from a single dose study will be analyzed at Day 1, Day 2, Day 30, Day 31, Day 150, and Day 180; multidose rollovers will just collect Day 1 and 180. Then there will be analyses every 6 months for 2.5 years, and annually for 3 years.
  Population and/or individual pharmacokinetic (PK) parameters for DCR PHXC, including maximum observed concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Verity Rawson, MB.CHB, Study Director — Dicerna, A Novo Nordisk Company
Locations (23):
- United States (4):
  - Clinical Research Site, San Francisco, California
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
- Australia (2):
  - Clinical Research Site, Herston, Queensland
  - Clinical Trial Site, Melbourne
- Clinical Research Site, Hamilton, Ontario, Canada
- France (2):
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Paris
- Germany (2):
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Heidelberg
- Clinical Research Site, Roma, Italy
- Japan (3):
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Nagoya
  - Clinical Trial Site, Tokyo
- Clinical Trial Site, Beirut, Lebanon
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, Tromsø, Norway
- Spain (2):
  - Clinical Research Site, Barcelona
  - Clinical Trial Site, Barcelona
- Clinical Trial Site, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Clinical Trial Site, Hampstead, London
  - Clinical Trial Site, Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Gamallo P, Rawson V. Population Pharmacokinetic and Pharmacodynamic Modelling and Simulation for Nedosiran Clinical Development and Dose Guidance in Pediatric Patients with Primary Hyperoxaluria Type 1. Clin Pharmacokinet. 2025 Sep;64(9):1395-1411. doi: 10.1007/s40262-025-01540-1. Epub 2025 Jul 2. PMID 40601241
- [Derived] Cox JH, Boily MO, Caron A, Sheng T, Wu J, Ding J, Gaudreault S, Chong O, Surendradoss J, Gomez R, Lester J, Dumais V, Li X, Gumpena R, Hall MD, Waterson AG, Stott G, Flint AJ, Moore WJ, Lowther WT, Knight J, Percival MD, Tong V, Oballa R, Powell DA, King AJ. Characterization of CHK-336, A First-in-Class, Liver-Targeted, Small-Molecule Lactate Dehydrogenase Inhibitor for Hyperoxaluria Treatment. J Am Soc Nephrol. 2025 Apr 7;36(8):1535-1547. doi: 10.1681/ASN.0000000690. PMID 40193200